CLINICAL TRIAL: NCT02995382
Title: Health-Related Quality of Life in Cases of Anterior Intramuscular Transposition for Cubital Tunnel Syndrome: A Prospective Cohort Study
Brief Title: Health-Related Quality of Life in Cases of Cubital Tunnel Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding was not received and the study could not proceed without this support.
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-2361
Record Dates: First submitted 2016-12-14; First posted 2016-12-16 (Estimated); Last update posted 2022-07-21 (Actual); Status verified 2021-09

CONDITIONS: Cubital Tunnel Syndrome
MeSH Terms: conditions — Cubital Tunnel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Anterior Intramuscular Transposition (Experimental): This is the only arm in our study, patients with cubital tunnel syndrome will undergo anterior intramuscular transposition, one of many surgical techniques utilized on patients with Cubital Tunnel Syndrome to alleviate symptoms.
  Interventions: Procedure: Anterior Intramuscular Transposition

INTERVENTIONS:
Procedure: Anterior Intramuscular Transposition — Anterior intramuscular transposition technique to decompress the ulnar nerve at the level of the elbow

SUMMARY:
This study aims to determine the Health Related Quality of life (HRQOL) (the physical, mental, emotional and social functioning) of patients with cubital tunnel syndrome following anterior intramuscular transposition, after one year.

DETAILED DESCRIPTION:
As there are many different surgical procedures to address cubital tunnel syndrome, HRQOL will be used to determine if anterior intramuscular transposition provides patients with positive outcomes. To measure HRQOL 3 specific scales will be administered:

1. A generic scale, the Short Form-36
2. A condition specific scale, the Patient-Rated Ulnar Nerve Evaluation (PRUNE)
3. A utility scale, the EuroQOL, five dimension questionnaire

These scales are widely reported in the literature, are valid, reliable and easy to fill out. Using these scales we can determine HRQOL as well as Quality Adjusted Life Years, which, allows us to do a cost-utility analysis (economic evaluation) on this specific procedure.

Patients will be asked to fill out the above mentioned questionnaires, as well as perform 2 performance tests (grip strength, and a moving 2-point discrimination test) at the following time points:

1. 1 week prior to surgery
2. 1 day prior to surgery
3. 3 months post surgery
4. 6 months post surgery
5. 12 months post surgery

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cubital tunnel syndrome confirmed with Electromyography (EMG) testing or Ultrasound imaging
* Ability to comprehend English and complete health related quality of life questionnaires
* Willing to provide informed consent
* Age > 18 years
* Not pregnant

Exclusion Criteria:

* Prior ipsilateral cubital tunnel release
* Evidence of symptomatic clinical double crush syndrome confirmed by EMG/Nerve Conduction Study (NCS)
* Patients with rheumatoid arthritis, connective tissue disorder, tenosynovitis, or diagnosed neurological condition that could confound the assessment of health-related quality of life with regard to the affected arm and hand

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Is there improvement in Health Related Quality of Life? | 1 week and 1 day pre-op & 3, 6, 12 months post op
  HRQOL will be determined using 3 questionnaires: a generic widely reported scale (SF-36), a condition specific valid and reliable scale (The PRUNE), and a utility scale EuroQol-5D)

SECONDARY OUTCOMES:
Which Domains of Health Related Quality of Life Improve? | 1 week and 1 day pre-op & 3, 6, 12 months post op
  There are different domains listed in the questionnaires, depending on the response from the patients we will determine where the improvement was seen (physical, mental, emotional, etc)
Is there improvement in physical performance? | 1 week and 1 day pre-op & 3, 6, 12 months post op
  This will be measured by using grip strength and moving 2-point discrimination

CONTACTS AND LOCATIONS:
Overall Officials: Matthew McRae, MD, Principal Investigator — McMaster University

IPD SHARING:
Plan to Share IPD: No
Data will not be shared to other researchers